CLINICAL TRIAL: NCT05944250
Title: A Pilot Study to Evaluate a Temporary Skin Substitute (Spincare® Matrix) for Wound Healing in RDEB Patients
Acronym: RDEB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean Yuh Tang, Professor of Dermatology, Stanford University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 69575
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Recessive Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Intervention Model Description: Intra-patient randomization of wound pairs into control wounds vs matrix treated wounds, followed by an open-label (extension) phase without randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Randomized Arm (Experimental): A full body wound examination will be performed by the investigator and target wound areas will be marked. All eligible wound sites will be randomized for matrix treatment versus standard of care wound dressings (at least 6 wounds, or 3 wound pairs). The matrix will be applied to randomized treatment wounds, along with a non-adhesive bandage as a protective layer.
  Interventions: Device: Spincare matrix
- Open-label Arm (extension) (Other): Participants who are eligible and choose to participate, will be enrolled at the 4 month long optional Open-Label Phase. Participant will be allowed to treat previously randomized wounds (treated and control wounds) and new wounds, up to a max of 10 individuals wounds; there won't be control or randomized wounds. Participants might reapply up to once a week, and wound healing and safety will be assessed at the monthly visits.
  Interventions: Device: Spincare matrix

INTERVENTIONS:
Device: Spincare matrix — The Spincare device, developed by Nanomedic, is the first portable tool that delivers a non-invasive, non-therapeutic electrospun, nanofibrous matrix dressing to wounds to promote healing.

SUMMARY:
Recessive dystrophic epidermolysis bullosa (RDEB) is a subtype of epidermolysis bullosa (EB), an inherited skin condition that presents with blistering skin. The Spincare device, developed by Nanomedic, is the first portable tool that delivers a non-invasive, non-therapeutic electrospun, nanofibrous matrix dressing to wounds to promote healing. The aim of this study is to determine the suitability of this device in RDEB wounds and assess its wound healing properties, safety and tolerability.

DETAILED DESCRIPTION:
Investigators will aim to recruit a mixture of adult and pediatric patient. However, the first patient that is recruited would be an adult to collect safety and efficacy data before enrolling pediatric patients.

Screening- Patients would be screened over the phone to assess if they meet the inclusion and exclusion criteria. Thereafter a virtual meeting via a secure virtual platform is arranged for the patient to review the consent form and sign. Wounds will be assessed to see if they meet the inclusion and exclusion criteria.

Day 0 - A full body wound examination will be performed by the investigator and target wound areas will be marked. All eligible wound sites will be randomized for matrix treatment versus standard of care wound care (at least 6 wounds, or 3 wound pairs). The matrix will be applied to randomized treatment wounds, along with a non-adhesive bandage as a protective layer. Reapplication of matrix treatment may be required depending on how well the matrix has propagated. At the time of matrix application, the investigator will score amount of wound burning, pain, or other adverse events. Non-treated wounds will have the patient's standard of care, non-adhesive bandage applied. Subjects and caregivers will be trained on how take photos. The aim is to capture photos of the wounds, pain and itch scores at least every 2 weeks. Surveys will be completed by the caregiver to see if they notice any difference in the wounds with the spray treatment. This will be completed together with the patient's pain and itch surveys.

Day 1 and optional Day 2- Clinic Visits: A wound examination will be performed in clinic. The investigator will assess the adherence of the matrix, and any adverse events (AEs). Day 2 visit may be necessary at the discretion of the investigators especially if any adverse events have occurred.

Months 1, 2, 3, 4 Visits: clinic attendance for patients with EB may be stressful and inconvenient due to their complex wound pattern and dressing changes. Keeping their safety and dignity as a priority the remaining visits as home visits are conducted with telehealth assessment. This will be done over a secure virtual platform or phone call whereby the assessors will be consulting remotely from a private Stanford based office room. The caregiver will apply the matrix to randomized, treated wounds (up to once a week application is allowed, the date and reason for reapplication is required)(additional interim visits/telehealth assessment and reapplication of matrix treatment may occur at Week 1, Week 2, Week 6, Week 10 and Week 14 or more frequently if deemed necessary). Patients will be asked to record the date each time the Spincare was applied. Photographs will be taken at those timepoints, and investigators will use Telehealth to monitor for healing and safety reporting (additional weekly photographs are encouraged). At the time of matrix application, the amount of wound burning, pain, or other adverse events will be scored Month 4 Telehealth/End of study Visit: The investigator will virtually assess wound healing compared to baseline photographs in the treated and control wounds. Digital photographs of the treatment and control wounds will be taken with a ruler by the caregiver and sent to the investigator. All wound photos will be reviewed via RedCAP. Wound swabs will be collected from treated and untreated wounds prior to spray treatment and at Month 2 and Month 4.

Participants may be offered the choice to complete surveys online and/or upload photos via Stanford RedCap.

Open-Label (Extension) Phase: After the completion of the 4-month randomized phase, patients will choose to enroll in an open Open-Label Phase for an additional 4 months. Investigators will conduct remote monitoring on a monthly basis to assess adverse events and wound healing. Participants will complete surveys regarding their pain and itch, offer updates on their medical history, and provide information about concurrent medications. No blood draws, wound cultures and in person visits will be required during the Open-Label Phase.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and/or genetic diagnosis of RDEB by a dermatologist
* Age 6 years or older willing and able to give consent/assent
* At least 6 wounds (3 wound pairs) each with an area of 10cm2 or greater located at any site (excluding face and genital skin)
* Wounds must be present for at least 4 weeks and able to be classified as recurrent wounds (wounds that heal within 12 weeks but then re-blister) vs chronic open (older than 12 weeks)

Exclusion Criteria:

* Actively infected wounds with pus (colonized wounds are eligible)
* Wounds that have had squamous cell carcinoma (SCC)
* Wounds on the face and genitals
* Wounds that have been treated with investigational therapies in the past 3 months

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Y Tang, PhD, Principal Investigator — Stanford University
Locations (1):
- Discovery Hall Stanford University, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified coded data may be shared with collaborators, funding agency and presented at scientific meetings. Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) would be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Immediately following publication. No end date
Access Criteria: Data will be presented at scientific meeting and in published material, Data may be available on sponsors website. Alternatively, proposals should be addressed to tangy@stanford.edu. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients aged 6-65 years with a clinical and/or genetic diagnosis of recessive dystrophic epidermolysis bullosa were screened over the phone. If eligible a virtual meeting was organized, and patients were asked to review and sign the informed consent form after which the wounds were assessed to determine suitability. This target population was chosen due to their large painful wounds usually resistant to conventional treatment and would benefit most from Spincare matrix treatment.
Pre-assignment Details: On Day 0, the investigator conducted an in-person full body skin examination and collected wound measurements to verify eligibility. The participant's wounds were assessed for signs of infection, and target wound areas were identified. Wounds that were actively infected with pus were excluded before randomization and the application of the matrix.
Units Other Than Participants: wounds
Groups:
- Matrix-Treated Wounds (Randomized Period); Standard of Care-Treated Wounds (Randomized Period): A full body wound examination was performed by the investigator and target wound areas were marked. All eligible wound sites were randomized for matrix treatment versus standard of care wound dressings (at least 6 wounds, or 3 wound pairs). The matrix was applied to randomized treatment wounds, along with a non-adhesive bandage as a protective layer.
- Open-label - Matrix Treatment: Participants from the randomized phase who were eligible and chose to participate, were enrolled at the 4 month long optional Open-Label Phase. Participant were allowed to treat previously randomized wounds (treated and control wounds) and new wounds, up to a max of 10 individuals wounds; there was no control or randomized wounds.
Period: Randomized Period (4 Months)
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period) | Open-label - Matrix Treatment
Started | 6; 21 wounds | 6; 21 wounds | 0; 0 wounds
Completed | 3; 11 wounds | 3; 11 wounds | 0; 0 wounds
Not Completed | 3; 10 wounds | 3; 10 wounds | 0; 0 wounds
Period: Open Label Period (4 Months)
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period) | Open-label - Matrix Treatment
Started | 0; 0 wounds | 0; 0 wounds | 1; 5 wounds
Completed | 0; 0 wounds | 0; 0 wounds | 1; 5 wounds
Not Completed | 0; 0 wounds | 0; 0 wounds | 0; 0 wounds

BASELINE CHARACTERISTICS:
Population: Patients aged 6 to 65 years old with a clinical and/or genetic diagnosis of recessive dystrophic epidermolysis bullosa. This is a pilot study in 6 subjects where wounds were randomized 1:1 to matrix application or no treatment (control).
Units Other Than Participants: wounds
Groups:
- Matrix-Treated Wounds (Randomized Period): Wounds that were randomized to receive matrix application.
- Standard of Care-Treated Wounds (Randomized Period): Wounds that were randomized to receive standard of care treatment.
- Open Label - Matrix-Treated: Wounds that were selected to receive matrix application, no randomization, no controls.
- Total: Total of all reporting groups
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period) | Open Label - Matrix-Treated | Total
Number analyzed (Participants) | 6 | 6 | 1 | 6
Number analyzed (wounds) | 21 | 21 | 5 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 0 | 4
  Between 18 and 65 years | 4 | 4 | 1 | 9
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 21 [11 to 32] | 21 [11 to 32] | 33 [33 to 33] | 21 [11 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 1 | 9
  Male | 2 | 2 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 0 | 6
  Not Hispanic or Latino | 2 | 2 | 1 | 5
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 1 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Wounds With Greater Than 90% Wound Closure at 4 Months
Description: The primary endpoint was comparison of the duration of wound closure of matrix-treated wounds vs control wounds measured as the number of wounds achieving greater than 90% wound closure within 4 months
Time Frame: Baseline to month 4 of the randomized phase
Population: Participants with month 4 data
Measure: Count of Units; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period)
Number analyzed (Participants) | 3 | 3
Number analyzed (Wounds) | 11 | 11
Wounds | 0 | 3
Statistical Analysis 1: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Test type: Superiority; p = 0.21, t-test, 2 sided

2. Secondary Outcome: Adverse Event Profile Characterization
Description: Comparison of application site adverse events (burning, erythema, pain) between matrix-treated wounds vs control wounds after application. For this outcome, adverse events were collected per wound; events affecting the participant but not the wound are not included.
Time Frame: 4-month randomized period followed by 4-month open-label period
Measure: Count of Units; unit: wounds
Units Other Than Participants: wounds
Groups:
- Matrix-Treated Wounds (Open Label Phase): A max. of 10 wounds per participant selected for matrix application. No controls, no randomization.
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period) | Matrix-Treated Wounds (Open Label Phase)
Number analyzed (Participants) | 6 | 6 | 1
Number analyzed (wounds) | 21 | 21 | 5
wounds
  Any Adverse Event | 11 | 10 | 0
  Pruritis, requiring medication to treat | 2 | 0 | 0
  Pain of Skin, requiring medication to treat | 3 | 0 | 0
  Bacterial Colonization | 0 | 4 | 0
  Skin Infection (non-serious) | 6 | 5 | 0

3. Secondary Outcome: Change From Baseline in Wound Pain Scale Score Assessment
Description: Pain was assessed using the Wong-Baker Faces scale (prior to matrix application). The scale consists of six faces that range from 0 (no pain at all, favorable outcome) to 10 (worst pain imaginable, worst outcome). Participants rated each wound using this scale, and scores were summed and averaged for each time point, resulting in an overall score range of 0 (no pain at all) to 10 (worst pain imaginable).
Time Frame: months 1, 2, 3, and 4 of the randomized phase
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: wounds
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period)
Number analyzed (Participants) | 6 | 6
Number analyzed (wounds) | 21 | 21
score on a scale
  Baseline | 3.143 (3.38) | 2.762 (3.71)
  Change at Month 1 | -1.43 (2.18) | -1.52 (3.64)
  Change at Month 2: number analyzed (Participants) | 4 | 4
  Change at Month 2: number analyzed (wounds) | 14 | 14
  Change at Month 2 | 0.43 (3.56) | -1.71 (3.42)
  Change at Month 3: number analyzed (Participants) | 3 | 3
  Change at Month 3: number analyzed (wounds) | 11 | 11
  Change at Month 3 | -1.45 (3.62) | -0.73 (4.96)
  Change at Month 4: number analyzed (Participants) | 3 | 3
  Change at Month 4: number analyzed (wounds) | 11 | 11
  Change at Month 4 | -1.64 (2.71) | -1.64 (3.8)

4. Secondary Outcome: Change in Wound Itch Scale Score Assessment
Description: Wound itch scores were assessed using the Itch NRS (prior to matrix application). The Itch NRS is a numerical rating scale from 0 to 10. Participants rated each wound using this scale, and scores were summed and averaged for each time point, resulting in an overall score of 0 to 10 (higher scores correspond to more pain).
Time Frame: months 1, 2, 3, and 4 of the randomized phase
Population: Participants with available data at the respective time point
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: wounds
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period)
Number analyzed (Participants) | 6 | 6
Number analyzed (wounds) | 21 | 21
units on a scale
  Baseline | 2.86 (2.55) | 2.10 (2.17)
  Change at Month 1 | -1.19 (1.24) | -0.71 (1.27)
  Change at Month 2: number analyzed (Participants) | 4 | 4
  Change at Month 2: number analyzed (wounds) | 14 | 14
  Change at Month 2 | -0.85 (2.75) | -0.43 (1.10)
  Change at Month 3: number analyzed (Participants) | 3 | 3
  Change at Month 3: number analyzed (wounds) | 11 | 11
  Change at Month 3 | -1.36 (1.55) | 0.27 (1.65)
  Change at Month 4: number analyzed (Participants) | 3 | 3
  Change at Month 4: number analyzed (wounds) | 11 | 11
  Change at Month 4 | -1.27 (1.59) | -0.18 (1.73)

5. Secondary Outcome: Number of Wounds That Reach >50% Healing From Baseline Per Investigator Assessment
Description: Comparison of wounds that reach >50% healing from baseline in matrix vs control (standard-of-care treated) wounds, per clinician assessment.
Time Frame: months 1, 2, 3, and 4 of the randomized phase
Population: Participants with available data at the respective time point
Measure: Number; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period)
Number analyzed (Participants) | 6 | 6
Number analyzed (Wounds) | 21 | 21
Wounds
  Month 1: number analyzed (Participants) | 5 | 5
  Month 1 | 8 | 7
  Month 2: number analyzed (Participants) | 4 | 4
  Month 2: number analyzed (Wounds) | 14 | 14
  Month 2 | 4 | 5
  Month 3: number analyzed (Participants) | 3 | 3
  Month 3: number analyzed (Wounds) | 11 | 11
  Month 3 | 4 | 4
  Month 4: number analyzed (Participants) | 3 | 3
  Month 4: number analyzed (Wounds) | 11 | 11
  Month 4 | 1 | 5
Statistical Analysis 1: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Wounds that reach >50% healing from baseline per investigator assessment at Month 1; Test type: Superiority; p = 1, t-test, 2 sided
Statistical Analysis 2: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Wounds that reach >50% healing from baseline per investigator assessment at Month 2; Test type: Superiority; p = 1, t-test, 2 sided
Statistical Analysis 3: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Wounds that reach >50% healing from baseline per investigator assessment at Month 3; Test type: Superiority; p = 1, t-test, 2 sided
Statistical Analysis 4: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Wounds that reach >50% healing from baseline per investigator assessment at Month 4; Test type: Superiority; p = 0.15, t-test, 2 sided

6. Secondary Outcome: Number of Wounds That Reach >70% Healing From Baseline Per Investigator Assessment
Description: Comparison of wounds that reach >70% healing from baseline in matrix-treated vs control wounds, per clinician assessment.
Time Frame: months 1, 2, 3, and 4 of the randomized phase
Population: Number of wounds that reach >70% healing from baseline in matrix-treated vs control wounds
Measure: Number; unit: Wounds
Units Other Than Participants: Wounds
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period)
Number analyzed (Participants) | 6 | 6
Number analyzed (Wounds) | 21 | 21
Wounds
  Month 1 | 4 | 5
  Month 2: number analyzed (Participants) | 4 | 4
  Month 2: number analyzed (Wounds) | 14 | 14
  Month 2 | 3 | 4
  Month 3: number analyzed (Participants) | 3 | 3
  Month 3: number analyzed (Wounds) | 11 | 11
  Month 3 | 1 | 3
  Month 4: number analyzed (Participants) | 3 | 3
  Month 4: number analyzed (Wounds) | 11 | 11
  Month 4 | 0 | 4
Statistical Analysis 1: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Wounds that reach >70% healing from baseline per investigator assessment at Month 1; Test type: Superiority; p = 1, t-test, 2 sided
Statistical Analysis 2: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Wounds that reach >70% healing from baseline per investigator assessment at Month 2; Test type: Superiority; p = 1, t-test, 2 sided
Statistical Analysis 3: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Wounds that reach >70% healing from baseline per investigator assessment at Month 3; Test type: Superiority; p = 0.59, t-test, 2 sided
Statistical Analysis 4: Comparison: Matrix-Treated Wounds (Randomized Period) vs Standard of Care-Treated Wounds (Randomized Period); Wounds that reach >70% healing from baseline per investigator assessment at Month 4; Test type: Superiority; p = 0.09, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4-month randomized period followed by 4-month open-label period
Groups:
- Matrix-Treated Wounds (Randomized Period): Adverse events localized to the area of the body with wounds that were randomized to receive matrix application.
- Standard of Care-Treated Wounds (Randomized Period): Adverse events localized to the area of the body with wounds that were randomized to receive standard of care treatment.
- Matrix-Treated Wounds (Open-Label Period): Adverse events localized to the area of the body with wounds that were selected to receive matrix application, no randomization, no controls.
- Systemic Adverse Events (Randomized Period); Systemic Adverse Events (Open-Label Period): All Adverse Events, including those that affected participants as a whole (systemic events)
Arm/Group | Matrix-Treated Wounds (Randomized Period) | Standard of Care-Treated Wounds (Randomized Period) | Matrix-Treated Wounds (Open-Label Period) | Systemic Adverse Events (Randomized Period) | Systemic Adverse Events (Open-Label Period)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/1 | 0/6 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/1 | 1/6 | 0/1
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 0/1 | 5/6 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Matrix-Treated Wounds (Randomized Period) (N=6) | Standard of Care-Treated Wounds (Randomized Period) (N=6) | Matrix-Treated Wounds (Open-Label Period) (N=1) | Systemic Adverse Events (Randomized Period) (N=6) | Systemic Adverse Events (Open-Label Period) (N=1)
Skin infection (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Cellulitis
Mammary Gland Carcinoma (Reproductive system and breast disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Invasive mammary gland neoplasm
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Matrix-Treated Wounds (Randomized Period) (N=6) | Standard of Care-Treated Wounds (Randomized Period) (N=6) | Matrix-Treated Wounds (Open-Label Period) (N=1) | Systemic Adverse Events (Randomized Period) (N=6) | Systemic Adverse Events (Open-Label Period) (N=1)
Fever (General disorders) | 0/0 | 0/0 | 0/0 | 1 | 0
Flu-like symptoms (Infections and infestations) | 0/0 | 0/0 | 0/0 | 3 | 0 — Unrelated to matrix treatment
Lymph node infection (Infections and infestations) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment
Headache, migraine (Nervous system disorders) | 0/0 | 0/0 | 0/0 | 0 | 1 — Unrelated to matrix treatment
Pruritis, requiring treatment (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 — Realted to matrix treatment
Pain of skin, requiring treatment (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 — Realted to matrix treatment
Bacterial colonization (Infections and infestations) | 0 | 2 | 0 | 2 | 0 — Unrelated to matrix treatment
Skin Infection (Infections and infestations) | 1 | 2 | 0 | 3 | 0 — Unrelated to matrix treatment
Toothache, chipped tooth (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment
Allergic reaction, seasonal allergies (Immune system disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment
Upper respiratory tract infection (Infections and infestations) | 0/0 | 0/0 | 0/0 | 2 | 0 — Unrelated to matrix treatment
Insomnia (Psychiatric disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment
Premature menopause (Reproductive system and breast disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment
Vaginal discharge (Reproductive system and breast disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment
Vision decreased, hyperopia (Eye disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment
Dental caries (Gastrointestinal disorders) | 0/0 | 0/0 | 0/0 | 1 | 0 — Unrelated to matrix treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT05944250/Prot_SAP_000.pdf